CLINICAL TRIAL: NCT04550416
Title: Effects of a New Diagnostic Test on the Care of Prostate Cancer Patients: The ProMark™ Clinical Utility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01-MM-14
Record Dates: First submitted 2014-06-13; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; risk assessment; clinical utility
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ProMark Information and Results (Experimental): Participants in the intervention arm will receive information (both print and webinar format) about ProMark in between Round 1 and Round 2 data collection, as well as appropriate ProMark test results for each of the vignette-based simulated patients that they care for in the second round of data collection.
  Interventions: Other: ProMark Information and Test Results
- Standard Practice (No Intervention): Physicians will care for online virtual patients as they normally would in practice.

INTERVENTIONS:
Other: ProMark Information and Test Results — Participants in the intervention arm will receive information (both print and webinar format) about ProMark in between Round 1 and Round 2 data collection, as well as appropriate ProMark test results for each of the vignette-based simulated patients that they care for in the second round of data collection.
  Arms: ProMark Information and Results

SUMMARY:
The objectives of this study are to assess clinical practice variation in prostate cancer diagnosis and treatment among urologists and how ProMark™ affects clinical practice decision-making. The study uses a randomized controlled study design of urologists. Urologists will be randomly assigned to a control and intervention arm.

* Pre-intervention/baseline assessment: will be done using prostate cancer CPV® vignettes and a physician questionnaire to both control and intervention arms.
* Intervention: 2-4 weeks after baseline introduce ProMark™ to the intervention group of urologists using a protocol to be determined by Metamark and QURE.
* Post-intervention: 6 weeks post-intervention, a second round of prostate cancer CPV® vignettes will be administered to both control and intervention arms. The ProMark™ test will be available to "order" for all physicians taking the vignettes.

The Clinical Performance and Value Vignettes (CPV®) used in this study simulate a clinical encounter for a man presenting with prostate cancer. Each urologist will provide responses to open-ended questions regarding clinical care they would provide for that patient. These responses are scored in five domains (taking a medical history, performing a physical examination, ordering appropriate tests, making a diagnosis and prescribing treatment against explicit evidence and criteria as determined by the literature and medical associations. Results are presented as percentage correct. Each case will take approximately 15-20 minutes to complete. All case responses will be completed online and kept confidential.

The study hypotheses are:

1. Clinical practice, specifically decisions around prostate cancer treatment post-diagnosis, will vary widely among urologists. This variation in practice will demonstrate the need a new diagnostic, such as ProMark™, would fulfill.
2. ProMark™ will improve clinical decision making of urologists for prostate cancer patients with a Gleason Score of 3+3=6 and 3+4=7 by improving the diagnosis and/or treatment CPV® domain score post-intervention versus baseline comparing intervention and control groups

The investigators will estimate the effect of ProMark™ on the primary outcomes comparing treatment and control groups using a difference-in-difference analysis comparing differences between groups before and after intervention. The investigators will control for potential confounders, such as age, gender, and other physician and practice characteristics.

DETAILED DESCRIPTION:
Secondary outcome measure include:

1. Difference in overall Clinical Performance and Value Vignettes (CPV®) scores post-intervention versus baseline comparing intervention and control groups
2. Difference between intervention and control for use of active surveillance.
3. Change in utilization of resources in terms of surgery, radiation (in any form), chemotherapy (in any of its forms) between intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Provide consent to participate in the study
* Currently practicing board certified urologist
* Have practiced as a board-certified urologist for greater than 2 or less than 30 years.
* English-speaking
* Community / non-academic based practice setting
* ≥50 PCa patients under care annually
* Access to the internet

Exclusion Criteria:

* Not board certified in urology
* Academic based practice
* Have previously used ProMark for prostate cancer care delivery
* Have practiced as a board-certified urologist for less than 2 or greater than 30 years.
* Follow <50 PCa patients annually
* Non-English speaking
* Unable to access the internet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Combined diagnostic and treatment CPV® (Clinical Performance and Value) vignette domain score | 12 to 16 weeks
  Difference in difference between the control and the intervention groups in the diagnosis-treatment quality of care as measured by their combined domain CPV scores (ranging from 0% to 100%) for the 9 patient types in aggregate and by case type.

CONTACTS AND LOCATIONS:
Overall Officials: John W Peabody, MD PhD, Principal Investigator — QURE Healthcare
Locations (1):
- QURE Healthcare, San Rafael, California, United States

REFERENCES:
- See also: Study Sponsor web page — http://www.metamarkgenetics.com